CLINICAL TRIAL: NCT00615290
Title: Pharmaco-epidemiological Description of the Patient Population Treated With Aptivus Under Market Conditions, Safety & Efficacy
Brief Title: Pharmaco-epidemiological Description of the Population Treated With Aptivus Under Market Conditions, Safety & Efficacy
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 1182.127
Record Dates: First submitted 2008-01-31; First posted 2008-02-14 (Estimated); Results first posted 2010-02-23 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — tipranavir

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Drug: tipranavir

SUMMARY:
To obtain information on clinical practices for patients treated by Aptivus in real life

ELIGIBILITY:
Inclusion Criteria:

* HIV positive patients for whom Aptivus treatment is initiated by their physician
* Aptivus SCP respect

Exclusion Criteria:

None if the inclusion criteria are respected: observational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2007-06; Primary Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (48):
- France (48):
  - Boehringer Ingelheim Investigational Site, Agen
  - Boehringer Ingelheim Investigational Site, Aix-en-Provence
  - Boehringer Ingelheim Investigational Site, Amiens
  - Boehringer Ingelheim Investigational Site, Argenteuil
  - Boehringer Ingelheim Investigational Site, Aulnay-sous-Bois
  - Boehringer Ingelheim Investigational Site, Auxerre
  - Boehringer Ingelheim Investigational Site, Belfort
  - Boehringer Ingelheim Investigational Site, Besançon
  - Boehringer Ingelheim Investigational Site, Béziers
  - Boehringer Ingelheim Investigational Site, Bondy
  - Boehringer Ingelheim Investigational Site, Bordeaux
  - Boehringer Ingelheim Investigational Site, Briis-sous-Forges
  - Boehringer Ingelheim Investigational Site, Cahors
  - Boehringer Ingelheim Investigational Site, Cannes
  - Boehringer Ingelheim Investigational Site, Chartres
  - Boehringer Ingelheim Investigational Site, Corbeil-Essonnes
  - Boehringer Ingelheim Investigational Site, Creil
  - Boehringer Ingelheim Investigational Site, Créteil
  - Boehringer Ingelheim Investigational Site, Dax
  - Boehringer Ingelheim Investigational Site, Digne-les-Bains
  - Boehringer Ingelheim Investigational Site, Garches
  - Boehringer Ingelheim Investigational Site, La Roche-sur-Yon
  - Boehringer Ingelheim Investigational Site, Le Mans
  - Boehringer Ingelheim Investigational Site, Le Petit-Quevilly
  - Boehringer Ingelheim Investigational Site, Libourne
  - Boehringer Ingelheim Investigational Site, Lyon
  - Boehringer Ingelheim Investigational Site, Mantes-la-Jolie
  - Boehringer Ingelheim Investigational Site, Marseille
  - Boehringer Ingelheim Investigational Site, Metz
  - Boehringer Ingelheim Investigational Site, Mulhouse
  - Boehringer Ingelheim Investigational Site, Nancy
  - Boehringer Ingelheim Investigational Site, Nantes
  - Boehringer Ingelheim Investigational Site, Nevers
  - Boehringer Ingelheim Investigational Site, Nice
  - Boehringer Ingelheim Investigational Site, Orléans
  - Boehringer Ingelheim Investigational Site, Paris
  - Boehringer Ingelheim Investigational Site, Périgueux
  - Boehringer Ingelheim Investigational Site, Poitiers
  - Boehringer Ingelheim Investigational Site, Rouen
  - Boehringer Ingelheim Investigational Site, Saint-Brieuc
  - Boehringer Ingelheim Investigational Site, Saint-Mandé
  - Boehringer Ingelheim Investigational Site, Saint-Nazaire
  - 1182.127.3301 Boehringer Ingelheim Investigational Site, Strasbourg
  - Boehringer Ingelheim Investigational Site, Strasbourg
  - Boehringer Ingelheim Investigational Site, Suresnes
  - Boehringer Ingelheim Investigational Site, Toulouse
  - Boehringer Ingelheim Investigational Site, Valenciennes
  - Boehringer Ingelheim Investigational Site, Villeneuve Saint G

RESULTS

PARTICIPANT FLOW:
Groups:
- Aptivus: Patients treated by Aptivus in daily practice
Period: Overall Study
Arm/Group | Aptivus
Started | 42
Completed | 34
Not Completed | 8
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: All enrolled patients
Arm/Group | Aptivus
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.9 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Viral Load< 50 Copies/mL and a Gain in CD4 Higher Than 100 Cells/mm3
Description: The evaluation at month 6 of an immunovirological response defined by a viral load less than 50 copies/mL and a gain in CD4 between day 0 and month 6 higher than 100 cells/mm3
Time Frame: 6 months after inclusion
Population: All enrolled patients with data at 6 months
Measure: Number; unit: participants
Arm/Group | Aptivus
Number analyzed (Participants) | 42
participants | 8

2. Secondary Outcome: Evaluation of Early Virological Response
Description: Number of patients presenting a decrease of viral load (HIV-RNA copies per mL) from day 0 to month 1 higher than 1 log10
Time Frame: 1 month after inclusion
Population: All enrolled patients with data at 1 month
Measure: Number; unit: participants
Arm/Group | Aptivus
Number analyzed (Participants) | 42
participants | 20

3. Secondary Outcome: Viral Load Response at 1 Month
Description: Please note that a reported value of "49 copies/mL" for the median or first quartile indicates that the observed statistic for the outcome measure is below the "limit of quantification" for viral load. The limit of quantification is 50 copies/mL.
Time Frame: 1 month after inclusion
Population: All enrolled patients with data at 1 month
Measure: Median (Inter-Quartile Range); unit: copies/mL
Arm/Group | Aptivus
Number analyzed (Participants) | 34
copies/mL | 71.5 [49 to 500]

4. Secondary Outcome: CD4 Count at 1 Month
Time Frame: 1 month after inclusion
Population: All enrolled patients with data at 1 month
Measure: Median (Inter-Quartile Range); unit: cells/cubic millimeter
Arm/Group | Aptivus
Number analyzed (Participants) | 35
cells/cubic millimeter | 349.0 [198.0 to 514.0]

5. Secondary Outcome: Evaluation of Intermediate Virological Response, Viral Load < 400 Copies/mL
Description: Number of patients with a viral load < 400 copies/mL after 3 months of treatment
Time Frame: 3 months after inclusion
Population: All enrolled patients with data at 3 months
Measure: Number; unit: participants
Arm/Group | Aptivus
Number analyzed (Participants) | 42
participants | 28

6. Secondary Outcome: Evaluation of Intermediate Virological Response, Viral Load < 50 Copies/mL
Description: Number of patients with a viral load < 50 copies/mL after 3 months of treatment
Time Frame: 3 months after inclusion
Population: All enrolled patients with data at 3 months
Measure: Number; unit: participants
Arm/Group | Aptivus
Number analyzed (Participants) | 42
participants | 24

7. Secondary Outcome: Viral Load Response at 3 Months
Description: as for outcome 3
Time Frame: 3 months after inclusion
Population: All enrolled patients with data at 3 months
Measure: Median (Inter-Quartile Range); unit: copies/mL
Arm/Group | Aptivus
Number analyzed (Participants) | 33
copies/mL | 49 [49 to 118]

8. Secondary Outcome: CD4 Count at 3 Months
Time Frame: 3 months after inclusion
Population: All enrolled patients with data at 3 months
Measure: Median (Inter-Quartile Range); unit: cells/cubic millimeter
Arm/Group | Aptivus
Number analyzed (Participants) | 34
cells/cubic millimeter | 322.5 [240.0 to 520.0]

9. Secondary Outcome: Patient Self Perception of the New Treatment
Description: Visual analogue scale range from 0 "not at all satisfied" to 100 "extremely satisfied"
Time Frame: Day 0, month 3 and month 6
Population: All enrolled patients
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Aptivus
Number analyzed (Participants) | 42
millimeter
  Day 0 (n=28) | 59 (25)
  Month 3 (n=28) | 76 (24)
  Month 6 (n=23) | 74 (25)

ADVERSE EVENTS:
Arm/Group | Aptivus
Serious Adverse Events (participants affected / at risk) | 3/42
Other Adverse Events (participants affected / at risk) | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aptivus (N=42)
Cytolitic hepatitis (Hepatobiliary disorders) | 2
Hepatitis (Hepatobiliary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.